CLINICAL TRIAL: NCT01915784
Title: Study Evaluating Preference, Satisfaction and Ease of Use of Genuair® (Pressair™) and Breezhaler® (Neohaler™) Inhalers in Chronic Obstructive Pulmonary Disease (COPD) Diagnosed Patients
Brief Title: Preference, Satisfaction and Ease of Use of Genuair® (Pressair™) and Breezhaler® (Neohaler™) Inhalers in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: M/34273/41
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Group A (Experimental): Genuair® (Pressair™) first; Breezhaler® (Neohaler™) second
  Interventions: Device: Genuair®; Device: Breezhaler®
- Group B (Experimental): Breezhaler® (Neohaler™) first; Genuair® (Pressair™) second
  Interventions: Device: Genuair®; Device: Breezhaler®

INTERVENTIONS:
Device: Genuair® — Inhaler with placebo only. Once daily, for 14 days.
  Other Names: Pressair™
Device: Breezhaler® — Inhaler with placebo only. Once daily, for 14 days.
  Other Names: Neohaler®

SUMMARY:
Preference study: Genuair® (Pressair™) vs Breezhaler® (Neohaler™) inhalers in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients aged ≥40 years with stable moderate-to-severe COPD according to the GOLD Guidelines classification (grades II and III): forced expiratory volume in 1 second (measured between 10 to 15 minutes post-inhalation of 400 μg of salbutamol) is 30%≤FEV1<80% of the predicted normal value
* Patients naïve to both study inhaler devices, Genuair® and Breezhaler®, for at least 2 years
* Agreement to participate and voluntarily sign the informed consent form

Exclusion Criteria:

* Patients with other clinically significant uncontrolled chronic diseases, particularly body malformations or diseases affecting coordination and/or motor system
* Patients unable to read product package instructions and answer patient reported questionnaires (PASAPQ)
* Patients with any other serious or uncontrolled mental health problems
* Patients currently participating in other randomised clinical studies
* Patients with COPD exacerbation within 6 weeks before Visit 1 and patient hospitalised for COPD exacerbation within 3 months prior to Visit 1
* Patients with any other conditions that, in the investigator's opinion, might indicate the patient to be inappropriate for the study
* Patient likely to be uncooperative

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who prefer Genuair® (Pressair™) versus Breezhaler® (Neohaler™) at Visit 2 | 14 Days
  Patients will be asked to answer which device they prefer after 2 weeks of daily practice recorded via PASAPQ (Patient Satisfaction and Preference Questionnaire) a self-administered, 15-item measure of respiratory inhalation device satisfaction and preference. The PASAPQ 15-item instrument includes 13 satisfaction items [using a Likert-type scale from 1 (very dissatisfied) to 7 (very satisfied)], a preference item, and a question on willingness to continue using the device.

SECONDARY OUTCOMES:
Mean for the overall satisfaction score with Genuair® (Pressair™) and Breezhaler® (Neohaler™) at Visit 2 | 14 Days
  Patients will be asked to rate the overall satisfaction with each device using a Likert-type scale (from 1 [very dissatisfied] to 7 [very satisfied]) after 2 weeks of daily practice recorded via PASAPQ (Patient Satisfaction and Preference Questionnaire) a self-administered, 15-item measure of respiratory inhalation device satisfaction and preference. The PASAPQ 15-item instrument includes 13 satisfaction items [using a Likert-type scale from 1 (very dissatisfied) to 7 (very satisfied)], a preference item, and a question on willingness to continue using the device.
Percentage of patients making at least 1 critical error with Genuair® (Pressair™) and Breezhaler® (Neohaler™) at Visit 2 | 14 Days
  The correct use of each device will be assessed measuring the errors made by patients when using each device after 2 weeks of daily practice
  Critical errors for each inhaler device are defined as those that compromise the potential benefit of the treatment such as impeding drug deposition in the lungs or the delivery of a sufficient dose

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Estruch, MD, Study Director — Almirall, S.A.
Locations (6):
- Germany (2):
  - Almirall investigative site 2, Berlin
  - Almirall investigative site 1, Munich
- Spain (2):
  - Almirall investigative site 3, Barcelona
  - Almirall investigative site 4, Palma de Mallorca
- United Kingdom (2):
  - Almirall investigative site 5, Glasgow
  - Almirall investigative site 6, Newcastle upon Tyne